CLINICAL TRIAL: NCT04018664
Title: A Study to Evaluate the Oral Abuse Potential of Nalbuphine Solution and Extended-Release Intact Tablets in Non-Dependent, Recreational Opioid Users
Brief Title: Oral Abuse Potential Study of Nalbuphine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: Protocol 1008910 (TR08)
Record Dates: First submitted 2019-05-30; First posted 2019-07-12 (Actual); Results first posted 2020-08-31 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Nalbuphine; Opioid Abuse
Keywords: nalbuphine; abuse potential
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Single-dose, randomized, double-blind, active- and placebo-controlled, double-dummy, 2-part, 7-way crossover study.
  Part A: Dose selection phase Part B: Treatment Periods 1-7
Who Masked: Participant, Care Provider, Investigator
Masking Description: For each dosing cohort, an unblinded statistician, not otherwise involved in the study, will prepare a list of subject randomization numbers. These randomization numbers will be used to prepare individual subject doses. Sealed qualification code break envelopes will be available for each subject in case of emergency.
  Upon completion of each cohort of subjects, the randomization codes for the completed subjects will be unblinded by the CRU pharmacy. After unblinding, the safety data will be reviewed to determine if dosing can proceed for the next planned dosing cohort,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Placebo (Placebo Comparator): Placebo
  150 mL flavored beverage
  Interventions: Drug: Placebo solution
- 90 mg nalbuphine HCl solution (Experimental): 90 mg nalbuphine HCl solution
  9 mL × 10 mg/mL hydromorphone HCl + 141 mL flavored beverage
  Interventions: Drug: Nalbuphine HCl solution
- 120 mg nalbuphine HCl solution (Experimental): 120 mg nalbuphine HCl solution
  12 mL × 10 mg/mL hydromorphone HCl + 138 mL flavored beverage
  Interventions: Drug: Nalbuphine HCl solution
- 150 mg nalbuphine HCl solution (Experimental): 150 mg nalbuphine HCl solution
  15 mL × 10 mg/mL hydromorphone HCl + 135 mL flavored beverage
  Interventions: Drug: Nalbuphine HCl solution
- 180 mg nalbuphine HCl solution (Experimental): 180 mg nalbuphine HCl solution
  18 mL × 10 mg/mL hydromorphone HCl + 132 mL flavored beverage
  Interventions: Drug: Nalbuphine HCl solution
- 270 mg nalbuphine HCl solution (Experimental): 270 mg nalbuphine HCl solution
  27 mL × 10 mg/mL hydromorphone HCl + 123 mL flavored beverage
  Interventions: Drug: Nalbuphine HCl solution
- Up to 405 mg nalbuphine HCl solution (Experimental): Up to 405 mg nalbuphine HCl solution
  Up to 40.5 mL × 10 mg/mL hydromorphone HCl + at least 109.5 mL flavored beverage
  Interventions: Drug: Nalbuphine HCl solution
- Up to 540 mg nalbuphine HCl solution (Experimental): Up to 540 mg nalbuphine HCl solution
  Up to 54 mL × 10 mg/mL hydromorphone HCl + at least 96 mL flavored beverage
  Interventions: Drug: Nalbuphine HCl solution

INTERVENTIONS:
Drug: Nalbuphine HCl solution — nalbuphine solution administered at various strengths
  Other Names: NAL ER
  Arms: 120 mg nalbuphine HCl solution; 150 mg nalbuphine HCl solution; 180 mg nalbuphine HCl solution; 270 mg nalbuphine HCl solution; 90 mg nalbuphine HCl solution; Up to 405 mg nalbuphine HCl solution; Up to 540 mg nalbuphine HCl solution
Drug: Placebo solution — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the effects of a drug called nalbuphine (an opioid drug) compared with the effects of hydromorphone (an opioid drug) and placebo (contains no active drug ingredients). The amount of nalbuphine levels in the blood will also be measured and the safety of the study drugs will be evaluated.

This study has 2 parts: Part A and Part B.

DETAILED DESCRIPTION:
This study will be a single-dose, randomized, double-blind, active- and placebo-controlled, double dummy, 2-part, 7-way crossover study to determine the abuse potential of orally administered nalbuphine solution and nalbuphine ER intact tablets relative to hydromorphone solution and placebo, in non-dependent, recreational opioid users. The study will be conducted in a single clinical research unit (CRU).

The purpose of Part A is to find the appropriate doses (a low, intermediate, and high dose) of nalbuphine solution to use in Part B. Part A of the study has two visits to the research clinic: a screening visit and dose selection visit. The visits will involve a 2-night stay (3 days total) in the research clinic.

In the Main Study Treatment Phase in Part B, the total estimated duration between each dose of study drug is approximately up to 7 days, of which the subject will spend 3 days/2 nights in the research clinic and approximately up to 4 days at home.

The primary objective of the Main Study is to evaluate the abuse potential of orally administered nalbuphine solution and nalbuphine ER intact tablets relative to hydromorphone solution (the active comparator) and placebo in non-dependent, recreational opioid users.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects 18 to 55 years of age
* Current opioid users who have used opioids for recreational (non-therapeutic) purposes

Exclusion Criteria:

* Self-reported substance or alcohol dependence (excluding nicotine and caffeine)
* Heavy smoker (≥ 20 cigarettes per day) and/or who is unable to abstain from smoking for at least 8 hours during the in clinic periods.
* History or presence of clinically significant abnormality as assessed by physical examination, medical history, ECGs, vital signs, or laboratory values.
* History or presence of any clinically significant illness
* History of major mental illness that may affect the ability of the subject to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2020-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics, Inc.
Locations (1):
- 001, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only Part A of this study was completed. Treatment arms summarized are those that were used on in Part A.
Groups:
- Placebo: Placebo
  150 mL flavored beverage
  Placebo solution: Placebo
- 90 mg Nalbuphine HCl Solution: 90 mg nalbuphine HCl solution
  9 mL × 10 mg/mL hydromorphone HCl + 141 mL flavored beverage
  Nalbuphine HCl solution: nalbuphine solution administered at various strengths
- 120 mg Nalbuphine HCl Solution: 120 mg nalbuphine HCl solution
  12 mL × 10 mg/mL hydromorphone HCl + 138 mL flavored beverage
  Nalbuphine HCl solution: nalbuphine solution administered at various strengths
- 150 mg Nalbuphine HCl Solution: 150 mg nalbuphine HCl solution
  15 mL × 10 mg/mL hydromorphone HCl + 135 mL flavored beverage
  Nalbuphine HCl solution: nalbuphine solution administered at various strengths
- 180 mg Nalbuphine HCl Solution: 180 mg nalbuphine HCl solution
  18 mL × 10 mg/mL hydromorphone HCl + 132 mL flavored beverage
  Nalbuphine HCl solution: nalbuphine solution administered at various strengths
- 270 mg Nalbuphine HCl Solution: 270 mg nalbuphine HCl solution
  27 mL × 10 mg/mL hydromorphone HCl + 123 mL flavored beverage
  Nalbuphine HCl solution: nalbuphine solution administered at various strengths
- Up to 405 mg Nalbuphine HCl Solution: Up to 405 mg nalbuphine HCl solution
  Up to 40.5 mL × 10 mg/mL hydromorphone HCl + at least 109.5 mL flavored beverage
  Nalbuphine HCl solution: nalbuphine solution administered at various strengths
- Up to 540 mg Nalbuphine HCl Solution: Up to 540 mg nalbuphine HCl solution
  Up to 54 mL × 10 mg/mL hydromorphone HCl + at least 96 mL flavored beverage
  Nalbuphine HCl solution: nalbuphine solution administered at various strengths
Period: Overall Study
Arm/Group | Placebo | 90 mg Nalbuphine HCl Solution | 120 mg Nalbuphine HCl Solution | 150 mg Nalbuphine HCl Solution | 180 mg Nalbuphine HCl Solution | 270 mg Nalbuphine HCl Solution | Up to 405 mg Nalbuphine HCl Solution | Up to 540 mg Nalbuphine HCl Solution
Started | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 90 mg Nalbuphine HCl Solution | 120 mg Nalbuphine HCl Solution | 150 mg Nalbuphine HCl Solution | 180 mg Nalbuphine HCl Solution | 270 mg Nalbuphine HCl Solution | Up to 405 mg Nalbuphine HCl Solution | Up to 540 mg Nalbuphine HCl Solution | Total
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (8.3) | 38.5 (11.2) | 33.2 (7.3) | 31.0 (9.4) | 37.3 (13.6) | 34.8 (5.6) | 34.3 (11.9) | 42.5 (12.3) | 35.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 8
  Male | 14 | 3 | 3 | 5 | 5 | 6 | 6 | 6 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 14 | 6 | 6 | 6 | 6 | 4 | 5 | 6 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 8
  White | 8 | 5 | 4 | 4 | 5 | 4 | 2 | 6 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 6
Region of Enrollment [Number; unit: participants]
  Canada | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56
BMI [Mean (Standard Deviation); unit: kg/m**2] | 26.48 (3.45) | 26.17 (3.15) | 25.53 (4.04) | 23.48 (2.57) | 26.18 (4.39) | 25.43 (3.62) | 24.53 (3.17) | 22.32 (1.55) | 25.23 (3.44)

OUTCOME MEASURES:

1. Primary Outcome: To Identify the Appropriate Low, Intermediarte, and High Doses of Nalbuphine Solution (Part A) to be Administered as Single Doses in the Treatment Phase of the Main Study (Part B).
Description: Only Part A of thie study was conducted because of closure the clinical research unit (CRU) before Part B could be initiated. Summary statistics are provided for C-max
Time Frame: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Population: C max
Measure: Mean (Standard Deviation); unit: microgram/L
Arm/Group | Placebo | 90 mg Nalbuphine HCl Solution | 120 mg Nalbuphine HCl Solution | 150 mg Nalbuphine HCl Solution | 180 mg Nalbuphine HCl Solution | 270 mg Nalbuphine HCl Solution | Up to 405 mg Nalbuphine HCl Solution | Up to 540 mg Nalbuphine HCl Solution
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 6
microgram/L |  | 21.70 (6.65) | 51.90 (26.89) | 68.67 (30.19) | 76.60 (51.34) | 56.00 (6.09) | 158.55 (115.65) | 196.83 (92.34)

ADVERSE EVENTS:
Time Frame: 24 days
Arm/Group | Placebo | 90 mg Nalbuphine HCl Solution | 120 mg Nalbuphine HCl Solution | 150 mg Nalbuphine HCl Solution | 180 mg Nalbuphine HCl Solution | 270 mg Nalbuphine HCl Solution | Up to 405 mg Nalbuphine HCl Solution | Up to 540 mg Nalbuphine HCl Solution
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT04018664/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT04018664/SAP_000.pdf